CLINICAL TRIAL: NCT05591339
Title: Diabetes Diagnosis, Management, Prevention and Education in Guinea-Bissau
Acronym: BCGTODM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: University of Coimbra (Other); Steno Diabetes Center Copenhagen (Other); University of Southern Denmark (Other); Sydvestjysk Sygehus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OP_1576
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus; BCG Vaccination Reaction
Keywords: BCG; Type-2 diabetes; non-specific effects; Guinea-Bissau
MeSH Terms: conditions — Diabetes Mellitus | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded to treatment. The investigators (or delegated vaccinator, e.g. nurse) administering the BCG vaccine or placebo (saline) will not be blinded. In case of serious adverse events, the participant can be unblinded after consultation with the coordinating PI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Experimental): Participants that are randomized in the active arm will receive an adult 0.1 ml dose of BCG vaccine (e.g. BCG-Denmark or BCG-Japan) in the skin covering the left upper deltoid muscle. Two doses will be given, 4 weeks apart.
  Intervention: Biological BCG-vaccine.
  Interventions: Biological: BCG vaccine (two doses, 4 weeks apart)
- Placebo (Placebo Comparator): Placebo will be 0.1 ml sterile 0.9 % NaCl, which has a similar color as the resuspended BCG vaccine. Two placebo doses will be given, 4 weeks apart.
  Interventions: Biological: Saline placebo (Two doses, 4 weeks apart)

INTERVENTIONS:
Biological: BCG vaccine (two doses, 4 weeks apart) — BCG vaccine provided intradermally at the upper arm.
  Arms: BCG vaccine
Biological: Saline placebo (Two doses, 4 weeks apart) — Participants randomized to the control group (placebo) will receive one 0.1 ml dose sterile 0.9 % NaCl by intradermal injection in the left deltoid region.
  Arms: Placebo

SUMMARY:
Type 2 diabetes (T2D) will affect ~650 million adults worldwide by 2040 and about as many will have pre-diabetes. Chronic hyperinsulinemia/insulin resistance precedes T2D development. Studies link insulin resistance with chronic inflammation and oxidative stress.

In Guinea-Bissau, a low-income country in West Africa, the T2D incidence is largely unknown and there is an acute lack of diabetes doctors, nurses and other diabetes educators. They hardly have access to insulin, and mortality from T2D complications is high. Previous studies by the Bandim Health Project (www.bandim.org) in the country show that the Bacillus Calmette-Guérin (BCG) vaccine has non-specific effects, well beyond tuberculosis prevention, conferring a general protection against unrelated pathogens. At the same time, studies from the US have also shown that BCG can significantly improve glycemic control in Type-1 diabetes (T1D) patients. Yet, no such studies have been done in T2D or pre-diabetes.

The purpose of the present study is to administer BCG to patients with pre-diabetes, in order to reduce hyperinsulinemia/chronic inflammation, a novel strategy to flatten the growing T2D incidence.

DETAILED DESCRIPTION:
BACKGROUND The lack of medical infrastructure and health education is clear across Guinea-Bissau, West Africa. Besides pilot studies from the capital Bissau, showing poor glycemic control and high mortality, due mainly to untreated type 2 diabetes (T2D), the diabetes prevalence is largely unknown. Patients cannot easily afford treatment, including insulin. Better health education, cheaper prevention and treatment strategies are needed.

Importantly, data show that the Bacillus Calmette Guerin (BCG) vaccine has key non-specific health effects, well beyond prevention of the target disease tuberculosis. Furthermore, in the US, it has been shown that BCG revaccination lowers haemoglobin-A1c (HbA1c) in people with Type-1 diabetes (T1D). Yet, no such studies have been done in T2D subjects.

The exact pathways of the non-specific effects of BCG are still being exploried, but it may be due to an increase in basal systemic levels of type 1 cytokines and immune cells and induction of epigenetic modifications in the innate immune cells, leading to increased pro-inflammatory responses towards unrelated pathogens. These modifications are accompanied by changes in glucose metabolism, increasing aerobic glycolysis, a state of high glucose utilization. In the randomized trial from the US in T1D patients, BCG lowered HbA1c close to normal levels. A systemic shift in glucose metabolism from oxidative phosphorylation to aerobic glycolysis was observed. BCG vaccination could therefore potentially be a cheap and safe tool to prevent T2D in resource-limited settings.

In Guinea-Bissau, only a couple of diabetes studies have been performed in patients with tuberculosis, HIV, twins and at a local diabetes clinic. Recently, study identified a severe lack of diabetes prevention, management and education. BCG vaccination could thus be a very valuable tool to prevent (and possibly treat) diabetes in low-income countries like Guinea-Bissau.

At the same time, studies indicate that long-term inflammation may predict dysmetabolism, independent of being lean or obese. Chronic inflammation is an important feature of insulin resistance and T2D, in which specific pro-inflammatory cytokines drive disease.

The rationale for the present study in Guinea-Bissau is therefore to test whether BCG vaccination could reduce HbA1c levels and ameliorate inflammation observed in individuals with pre-diabetes, thereby preventing the progression to overt T2D.

AIM OF STUDY Conduct a randomized trial to investigate the metabolic effects of two BCG vaccinations 4 weeks apart in persons with pre-diabetes. Metabolic status is monitored during the trial and related with inflammatory biomarkers.

MAIN HYPOTHESIS Providing two BCG vaccinations 4 weeks apart to individuals with pre-diabetes, compared with placebo, is associated with lower fasting glucose/hba1c levels at 3 years follow-up.

DEFINITIONS Pre-diabetes: F-glucose between 5.6-6.9 mmol/L or HbA1c between 39-47mmol/L. Above these levels is diabetes.

INVESTIGATIONS AND SAMPLE SIZE

The aim is to conduct a randomized trial to investigate the metabolic effects of two BCG vaccinations 4 weeks apart in pre-diabetes adult subjects. The pre-diabetes patients will partly be identified in a diabetes prevalence study being conducted prior to the trial.

The participants are followed for 3 consecutive years, with F-glucose and hba1c measured every 3 months.

Metabolic status is monitored by measuring metabolic markers (glucose, hba1c, insulin, leptin, adiponectin) and relating these with inflammatory markers (Il-6, Il-10, Il-33, TNFa) pre and post-trial.

The blood for the advanced metabolic and inflammatory biomarkers will be collected and stored in frozen condition (-40C) in Guinea-Bissau at the National Health Laboratory (LNSP), before being transported to Coimbra University, Portugal, for analyses.

Sample size: If anticipating at 3 years follow-up a reduction in mean F-glucose from 7.0 mmol/L to 6.0, there would be a need 63 participants in each group, with a potency of 80% and an alpha of 0.05. Therefore, including a total of 200 participants with pre-diabetes in this BCG study should give us an appropriate sample size, also taking into account loss to follow-up.

SETTING The trial will be conducted by the Bandim Health Project (BHP) team in Bissau (www.bandim.org). Since 1978, the BHP has maintained a health and demographic surveillance system (HDSS) site here.

The National Diabetes Clinic (NDC): Is the only diabetes clinic in Guinea-Bissau, situated within the BHP study area, where the trial will take place. The clinic is semi-private and run by the Guinean Diabetes Association (ANDD).

METHODS The investigators will invite 200 individuals with pre-diabetes. Provided the participants meets the inclusion/exclusion criteria, fasting blood samples will be collected by a team nurse. Clinical records will contain demographic characteristics, patient history, anthropometry, clinical measurements, prescriptions, diagnoses and the presence of diabetic wounds. BCG and smallpox vaccination scar status are assessed.

Follow-up: Participants will be recalled for evaluation every three months, during the 3 years trial, where the investigators will measure F-glucose and HbA1c levels.

Glycemic analyses: F-glucose levels will be measured using Accu-Chek Aviva. Hb1Ac will be measured on a Bayer's A1CNow.

Bio markers: At baseline and every 6 months during follow-up the investigators will measure metabolic (glucose, hba1c, insulin, leptin, adiponectin) and inflammatory markers (Il-6, Il-10, Il-33, TNFa).

Data management: After randomization, the participants will receive a card with a unique study number, which they need to bring to facilitate identification. All information will be entered in RedCap.

STATISTICS BCG's effect on F-glucose and hba1c will be done using Poisson regression models, and time to T2D diagnosis by Cox regression. Analyses will be done overall, by sex and pre-diabetes levels. It will be examined whether prior BCG-scaring affects the intervention.

ETHICAL CONSIDERATIONS The protocol has been approved by to the Guinean Ethical Committees. Informed written consent will be obtained before enrolment.

DATA SAFETY AND MONITORING BOARD This will be established consisting of a diabetes expert and a statistician plus an additional member.

NOVELTY AND SIGNIFICANCE Better diabetes prevention and treatment strategies are urgently needed. If the trial is successful, it will represent a major improvement in the diabetes control, and at very low cost. Essentially, with the proper handling techniques, BCG can be administered everywhere, even in the most resource-limited areas.

SPONSOR: The BHP and the University of Coimbra (UC) are both the sponsors of the study, and wrote the protocol jointly. The UC is therefore also a co-responsible party.

ELIGIBILITY:
Inclusion Criteria for BCG trial:

* Ages 18-64
* Planning to continue living in the study area
* F-glucose from 5.6-6.9 mmol/L and HbA1c between 39-47mmol/mol.

Exclusion Criteria for BCG trial:

* HIV infection (an HIV test to be done before enrolment)
* Pregnancy (a pregnancy test to be done before enrolment in women in the childbearing age)
* Chemotherapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Hba1c | 3 years after enrolment
  Hba1c levels at the end of the study period in people with pre-diabetes
F-glucose | 3 years after enrolment
  F-glucose levels at the end of the study period in people with pre-diabetes

SECONDARY OUTCOMES:
Type-2 diabetes | 3 years after enrolment
  Confirmed Type-2 diabetes at the end of the study period in people with pre-diabetes
Time to Type-2 diabetes development | 0-3 years after enrolment
  Number of months between enrolment and development of Type-2 diabetes in people with pre-diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Carvalho, PhD, Study Chair — Center of Neuroscience and Cell Biology, University of Coimbra, Portugal; Lilica Sanca, Bsc, Principal Investigator — Bandim Health Project; Morten Bjerregaard-Andersen, MD, PhD, Principal Investigator — Hospital of Southwest Jutland, Denmark; Stine Byberg, MSc, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data can be shared after approval of a data-sharing proposal submitted to the study chair person (Eugenia Carvalho).

REFERENCES:
- [Background] Correia JC, Lopes A, Iala CB, Sanca NA, Bidonga A, Lagger G, Golay A, Castellsague MP. Diabetes management in Guinea Bissau: a situational analysis. Pan Afr Med J. 2019 Sep 4;34:10. doi: 10.11604/pamj.2019.34.10.19874. eCollection 2019. PMID 31762879
- [Background] Byberg S, Bundesen C, Rudolf F, Haraldsdottir TL, Indjai L, Barai R, Beck-Nielsen H, Sodemann M, Jensen DM, Bjerregaard-Andersen M. Diabetes in urban Guinea-Bissau; patient characteristics, mortality and prevalence of undiagnosed dysglycemia. Glob Health Action. 2020 Dec 31;13(1):1802136. doi: 10.1080/16549716.2020.1802136. PMID 32814520
- [Background] Benn CS, Roth A, Garly ML, Fisker AB, Schaltz-Buchholzer F, Timmermann A, Berendsen M, Aaby P. BCG scarring and improved child survival: a combined analysis of studies of BCG scarring. J Intern Med. 2020 Dec;288(6):614-624. doi: 10.1111/joim.13084. Epub 2020 May 25. PMID 32301189
- [Background] Schaltz-Buchholzer F, Aaby P, Monteiro I, Camala L, Faurholt Simonsen S, Nortoft Frankel H, Lindberg Larsen K, Golding CN, Kollmann TR, Amenyogbe N, Stabell Benn C, Bjerregaard-Andersen M. Immediate Bacille Calmette-Guerin Vaccination to Neonates Requiring Perinatal Treatment at the Maternity Ward in Guinea-Bissau: A Randomized Controlled Trial. J Infect Dis. 2021 Dec 1;224(11):1935-1944. doi: 10.1093/infdis/jiab220. PMID 33893799
- [Background] Aaby P, Benn CS. BCG: new life for a centenarian vaccine. Lancet Infect Dis. 2021 Jul;21(7):897-898. doi: 10.1016/S1473-3099(20)30714-3. Epub 2021 Feb 17. No abstract available. PMID 33609459
- [Background] Kuhtreiber WM, Tran L, Kim T, Dybala M, Nguyen B, Plager S, Huang D, Janes S, Defusco A, Baum D, Zheng H, Faustman DL. Long-term reduction in hyperglycemia in advanced type 1 diabetes: the value of induced aerobic glycolysis with BCG vaccinations. NPJ Vaccines. 2018 Jun 21;3:23. doi: 10.1038/s41541-018-0062-8. eCollection 2018. PMID 29951281
- [Background] Faustman DL, Wang L, Okubo Y, Burger D, Ban L, Man G, Zheng H, Schoenfeld D, Pompei R, Avruch J, Nathan DM. Proof-of-concept, randomized, controlled clinical trial of Bacillus-Calmette-Guerin for treatment of long-term type 1 diabetes. PLoS One. 2012;7(8):e41756. doi: 10.1371/journal.pone.0041756. Epub 2012 Aug 8. PMID 22905105
- [Background] Biering-Sorensen S, Jensen KJ, Monterio I, Ravn H, Aaby P, Benn CS. Rapid Protective Effects of Early BCG on Neonatal Mortality Among Low Birth Weight Boys: Observations From Randomized Trials. J Infect Dis. 2018 Feb 14;217(5):759-766. doi: 10.1093/infdis/jix612. PMID 29216358
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Mbanya JC, Motala AA, Sobngwi E, Assah FK, Enoru ST. Diabetes in sub-Saharan Africa. Lancet. 2010 Jun 26;375(9733):2254-66. doi: 10.1016/S0140-6736(10)60550-8. PMID 20609971
- [Background] Meiloud G, Arfa I, Kefi R, Abdelhamid I, Veten F, Lasram K, Ben Halim N, Sidi Mhamed A, Samb A, Abdelhak S, Houmeida AO. Type 2 diabetes in Mauritania: prevalence of the undiagnosed diabetes, influence of family history and maternal effect. Prim Care Diabetes. 2013 Apr;7(1):19-24. doi: 10.1016/j.pcd.2012.12.002. Epub 2013 Feb 4. PMID 23380050
- [Background] Bjerregaard-Andersen M, Hansen L, da Silva LI, Joaquim LC, Hennild DE, Christiansen L, Aaby P, Benn CS, Christensen K, Sodemann M, Jensen DM, Beck-Nielsen H. Risk of metabolic syndrome and diabetes among young twins and singletons in Guinea-Bissau. Diabetes Care. 2013 Nov;36(11):3549-56. doi: 10.2337/dc12-2653. Epub 2013 Aug 15. PMID 23949562
- [Background] Haraldsdottir TL, Rudolf F, Bjerregaard-Andersen M, Joaquim LC, Stochholm K, Gomes VF, Beck-Nielsen H, Ostergaard L, Aaby P, Wejse C. Diabetes mellitus prevalence in tuberculosis patients and the background population in Guinea-Bissau: a disease burden study from the capital Bissau. Trans R Soc Trop Med Hyg. 2015 Jun;109(6):400-7. doi: 10.1093/trstmh/trv030. Epub 2015 Apr 26. PMID 25918218
- [Background] Steiniche D, Jespersen S, Erikstrup C, Krarup H, Handberg A, Ostergaard L, Haraldsdottir T, Medina C, Gomes Correira F, Laursen AL, Bjerregaard-Andersen M, Wejse C, Honge BL; Bissau HIV Cohort study group. Diabetes mellitus and impaired fasting glucose in ART-naive patients with HIV-1, HIV-2 and HIV-1/2 dual infection in Guinea-Bissau: a cross-sectional study. Trans R Soc Trop Med Hyg. 2016 Apr;110(4):219-27. doi: 10.1093/trstmh/trw017. PMID 27076509
- [Background] Fischer IP, Irmler M, Meyer CW, Sachs SJ, Neff F, Hrabe de Angelis M, Beckers J, Tschop MH, Hofmann SM, Ussar S. A history of obesity leaves an inflammatory fingerprint in liver and adipose tissue. Int J Obes (Lond). 2018 Mar;42(3):507-517. doi: 10.1038/ijo.2017.224. Epub 2017 Sep 13. PMID 28901330
- [Background] Denis GV, Obin MS. 'Metabolically healthy obesity': origins and implications. Mol Aspects Med. 2013 Feb;34(1):59-70. doi: 10.1016/j.mam.2012.10.004. Epub 2012 Oct 13. PMID 23068072
- [Background] DeFuria J, Belkina AC, Jagannathan-Bogdan M, Snyder-Cappione J, Carr JD, Nersesova YR, Markham D, Strissel KJ, Watkins AA, Zhu M, Allen J, Bouchard J, Toraldo G, Jasuja R, Obin MS, McDonnell ME, Apovian C, Denis GV, Nikolajczyk BS. B cells promote inflammation in obesity and type 2 diabetes through regulation of T-cell function and an inflammatory cytokine profile. Proc Natl Acad Sci U S A. 2013 Mar 26;110(13):5133-8. doi: 10.1073/pnas.1215840110. Epub 2013 Mar 11. PMID 23479618
- [Background] Denis GV, Sebastiani P, Bertrand KA, Strissel KJ, Tran AH, Slama J, Medina ND, Andrieu G, Palmer JR. Inflammatory signatures distinguish metabolic health in African American women with obesity. PLoS One. 2018 May 8;13(5):e0196755. doi: 10.1371/journal.pone.0196755. eCollection 2018. PMID 29738558
- [Background] Bastard JP, Maachi M, Lagathu C, Kim MJ, Caron M, Vidal H, Capeau J, Feve B. Recent advances in the relationship between obesity, inflammation, and insulin resistance. Eur Cytokine Netw. 2006 Mar;17(1):4-12. PMID 16613757
- [Background] Hennild DE, Bjerregaard-Andersen M, Joaquim LC, Christensen K, Sodemann M, Beck-Nielsen H, Jensen DM. Prevalence of impaired glucose tolerance and other types of dysglycaemia among young twins and singletons in Guinea-Bissau. BMC Endocr Disord. 2016 Aug 4;16(1):46. doi: 10.1186/s12902-016-0126-6. PMID 27491662
- [Background] Awah PK, Unwin NC, Phillimore PR. Diabetes Mellitus: Indigenous naming, indigenous diagnosis and self-management in an African setting: the example from Cameroon. BMC Endocr Disord. 2009 Feb 19;9:5. doi: 10.1186/1472-6823-9-5. PMID 19224650
- [Background] Abdulrehman MS, Woith W, Jenkins S, Kossman S, Hunter GL. Exploring Cultural Influences of Self-Management of Diabetes in Coastal Kenya: An Ethnography. Glob Qual Nurs Res. 2016 Apr 8;3:2333393616641825. doi: 10.1177/2333393616641825. eCollection 2016 Jan-Dec. PMID 28462335
- See also: Bandim Health Project in Guinea-Bissau — http://www.bandim.org